CLINICAL TRIAL: NCT05534139
Title: Clinicopathological MRI and CSF Correlates of Iron Accumulation, Neurodegeneration and Neuroinflammation in Huntington's Disease.
Brief Title: Clinicopathological MRI and CSF Correlates in Huntington's Disease.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Brighton & Sussex Medical School (Other); University of Ulm (Other)
Responsible Party: Principal Investigator, Susanne T de Bot, MD, PhD, MD PhD, Leiden University Medical Center
Other Study IDs: P19.030
Record Dates: First submitted 2022-08-15; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Huntington Disease
Keywords: Huntington's Disease; Iron accumulation; Quantified susceptibility mapping; QSM; 7T-MRI; CSF; Neurodegeneration; Neuroinflammation
MeSH Terms: conditions — Huntington Disease; Nerve Degeneration; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood and CSF (collected in a fasted state)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy controls: Partner/spouse of a patient not at risk of HD OR sibling with genetic test results available that show a normal CAG repeat length for both HTT alleles (<36); No other known cognitive, neurological or psychiatric disorders.
  Interventions: Diagnostic Test: 7T MRI-scan; Diagnostic Test: CSF collection via lumbar puncture; Diagnostic Test: Blood withdrawal; Diagnostic Test: Clinical measures
- Premanifest HD expanded gene carrier: HDGEC before clinical onset: TMS <5, DCL <4, TFC = 13. No other major comorbidity.
  Interventions: Diagnostic Test: 7T MRI-scan; Diagnostic Test: CSF collection via lumbar puncture; Diagnostic Test: Blood withdrawal; Diagnostic Test: Clinical measures
- Early Manifest HD patient: HDGEC after clincial onset: TMS >5, DCL = 4. Early stage of disease: TFC 11-13. No other major comorbidity.
  Interventions: Diagnostic Test: 7T MRI-scan; Diagnostic Test: CSF collection via lumbar puncture; Diagnostic Test: Blood withdrawal; Diagnostic Test: Clinical measures
- Moderate Manifest HD patient: HDGEC after clincial onset: TMS >5, DCL = 4. Moderate stage of disease: TFC 7-10. No other major comorbidity.
  Interventions: Diagnostic Test: 7T MRI-scan; Diagnostic Test: CSF collection via lumbar puncture; Diagnostic Test: Blood withdrawal; Diagnostic Test: Clinical measures

INTERVENTIONS:
Diagnostic Test: 7T MRI-scan — MRI-scanning of the brain using a 7T-MRI scanner
Diagnostic Test: CSF collection via lumbar puncture — CSF is collected by doing a lumbar puncture
Diagnostic Test: Blood withdrawal — Blood is collected by doing a blood withdrawal
Diagnostic Test: Clinical measures — UHDRS-Total motor score, UHDRS-short problem behaviour assessment, UHDRS-Cognitive assessments

SUMMARY:
In this study the investigators will link brain iron levels obtained from quantitative susceptibility maps of HD patients with specific and well-known clinical CSF markers for iron accumulation, neurodegeneration and neuroinflammation. The relationship between iron accumulation and neuroinflammation, and the clinical and genetic characteristics of HD will be investigated. This will provide an important basis for the evaluation of brain iron levels as an imaging biomarker for disease state in HD and their relationship with the salient pathomechanisms of the disease.

DETAILED DESCRIPTION:
This investigator-initiated, single-site cross-sectional study looks at iron accumulation using 7T MR-imaging, CSF and blood. This will be achieved in a two-day visit involving clinical assessments, MRI-scanning of the brain, followed by a lumbar puncture the next day, after overnight fasting. Sixty-five volunteers with HD and 25 volunteers without HD will be included. Of these 65 volunteers with HD, 25 will be premanifest, 20 early manifest and 20 moderate manifest, in order to cover the wide-spectrum of Huntington's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Native Dutch/Flemish speaker
* Ability to undergo MRI scanning;
* Written informed consent must be obtained from the participant.

And in addition:

If the participant is a pre-manifest HD gene carrier:

* CAG expansion ≥ 40;
* UHDRS Total Motor Score (TMS) ≤ 5;
* Total Functional Capacity (TFC) = 13;
* Diagnostic Confidence Score < 4.

If the participant is an early-manifest HD gene carrier:

* CAG expansion ≥ 36;
* Diagnostic Confidence Score = 4;
* HD stage I: TFC scores between 11 and 13 inclusive.

If the participant is a moderate manifest HD gene carrier:

* CAG expansion ≥ 36;
* Diagnostic Confidence Score = 4;
* HD stage II: TFC scores between 7 and 11 inclusive.

If the participant is a control subject:

* Partner/spouse of a patient not at risk of HD OR sibling with genetic test results available that show a normal CAG repeat length for both HTT alleles (<36);
* No other known cognitive, neurological or psychiatric disorders.

Exclusion Criteria:

* Additional major comorbidities not related to HD (e.g. cardiovascular diseases, coagulopathy, hypertension, diabetes mellitus, and/or other neurological disorders);
* History of severe head injury;
* Status of the participant after brain surgery;
* Past erythrocyte transfusions;
* Use of investigational drugs or participation in a clinical drug trial within 30 days prior to study visit;
* Current intoxication, drug or alcohol abuse or dependence;
* Pregnancy;
* Inability to understand the information about the protocol;
* Severe physical restrictions (completely wheelchair dependent);
* Severe chorea that, in the investigator's judgment, precludes the patient's participation in and completion of the MRI and/or lumbar puncture.
* Contra-indication to MRI scanning, such as:

  * Claustrophobia;
  * Pacemakers and defibrillators;
  * Nerve stimulators;
  * Intracranial clips;
  * Intraorbital or intraocular metallic fragments;
  * Cochlear implants;
  * Ferromagnetic implants;
  * Hydrocephalus pump;
  * Intra-utrine device (not all types);
  * Permanent make-up;
  * Tattoos above the shoulders (not all).
* Contraindications for a lumbar puncture, including:

  * Screening blood test results outside normal ranges(white cell count, neutrophil count, lymphocyte count, hemoglobin, platelets, Prothrombin time (PT), activated partial thromboplastin time (APTT), C-reactive protein (CRP) and serum ferritin) if only marginally decreased or increased this will be decided by the clinical PI;
  * Signs and symptoms of increased intracranial pressure which will be confirmed on the 7T MRI (T1 and FLAIR scan) or by a fundoscopy;
  * Local infections of the skin;
  * Use of anti-coagulant drugs within the last 14 days prior lumbar puncture.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pre-manifest HD gene carrier:
  * CAG expansion ≥ 40;
  * UHDRS Total Motor Score (TMS) ≤ 5;
  * Total Functional Capacity (TFC) = 13;
  * Diagnostic Confidence Score < 4.
  Early-manifest HD gene carrier:
  * CAG expansion ≥ 36;
  * Diagnostic Confidence Score = 4;
  * HD stage I: TFC scores between 11 and 13 inclusive.
  Moderate manifest HD gene carrier:
  * CAG expansion ≥ 36;
  * Diagnostic Confidence Score = 4;
  * HD stage II: TFC scores between 7 and 10
  Control subject:
  * Partner/spouse of a patient not at risk of HD OR sibling with genetic test results available that show a normal CAG repeat length for both HTT alleles (<36);
  * No other known cognitive, neurological or psychiatric disorders.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Quantified Susceptibility Mapping | At baseline
  MRI analysis to quantify iron accumulation
Iron in CSF | At baseline
  Amount of iron and ferritin measured in CSF

SECONDARY OUTCOMES:
Iron in blood | At baseline
  Amount of iron and ferritin measured in blood
Clinical motor signs | At baseline
  Motor signs obtained using the Unified Huntington's Disease Rating Scale - Total Motor Score. This is a scale assessing motor symptoms of HD, ranging from a score of 0 to 124, where higher scores mean a worse outcome.
Neuroinflammation and neurodegeneration biomarkers in CSF | Baseline
  a.o.
  * NFL: pg/mL
  * CHIT1: pg/mL
  * IL-6: pg/mL
Neuroinflammation and neurodegeneration biomarkers in CSF | Baseline
  - YKL-40: ng/mL
Cognitive score | At baseline
  Assessment of cognitive tests.
Neuropsychiatric symptoms | At baseline
  Assessment of short Problem Behaviour Assessment. Each symptom is rated for severity on a 5-point scale : 0 = "not at all"; 1 = trivial; 2 = mild; 3 = moderate (disrupting everyday activities) and 4 = severe or intolerable. Each symptom is also scored for frequency on a 5-point scale as follows: 0 = symptom absent; 1 = less than once weekly; 2 = at least once a week; 3 = most days (up to and including some part of everyday); and 4 = all day, every day. Severity and frequency scores are multiplied to produce an overall 'PBA score' for each symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne de Bot, MD PhD, Principal Investigator — Neurology
Locations (1):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No